CLINICAL TRIAL: NCT01558661
Title: A Phase II Study of Axitinib (AG-013736) in Patients With Progressive, Recurrent/Metastatic Adenoid Cystic Carcinoma
Brief Title: Axitinib (AG-013736) in Patients With Progressive, Recurrent/Metastatic Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-004
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2016-08

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: axitinib (AG-013736); recurrent; metastatic; 12-004
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Recurrence; Neoplasm Metastasis | interventions — Axitinib

ARMS (1):
- AG-013736 (AXITINIB) (Experimental): This is a single-arm phase II study evaluating the clinical efficacy of axitinib in the treatment of patients with progressive, recurrent/metastatic adenoid cystic carcinoma (ACC).
  Interventions: Drug: AG-013736 (AXITINIB)

INTERVENTIONS:
Drug: AG-013736 (AXITINIB) — All eligible patients will receive a starting axitinib dose of 5 mg twice daily (BID) taken orally in 4-week (28-day) cycles. Patients who tolerate axitinib with no adverse events related to study drug above CTCAE v. 4.0 Grade 2 for a consecutive 2-week period may have their dose increased by one dose level according to the discretion of the treating physician (NOT allowed for patients with blood pressure (BP) > 150/90 mm Hg or who are receiving antihypertensive medication). This dose escalation is not mandatory. RECIST v1.1 tumor assessments will be made at baseline (CT or MRI) and then approximately every 2 cycles (or every 8 weeks (+/- 1 week)). After 10 months, imaging will be done every 3 cycles (or every 12 weeks (+/- 1 week)). Patients may remain on study until progression of disease or unacceptable toxicity.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, a new treatment called axitinib has on the patient and adenoid cystic carcinoma. This type of cancer study is called a phase II study.

Axitinib is an oral medication that can interfere with cancer cell growth and reduce the growth of blood vessels around tumors. This study will help find out if axitinib is a useful drug for treating patients with adenoid cystic carcinomas. Axitinib is an experimental drug that has not yet been approved by the Food and Drug Administration for use in adenoid cystic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have MSKCC pathologically confirmed adenoid cystic carcinoma. Cancers arising from non-salivary gland primary sites are allowed.
* Patients must have locally advanced and/or recurrent and/or metastatic disease not amenable to potentially curative surgery or radiotherapy.
* At least 2 weeks must have elapsed since the end of prior systemic treatment (4 weeks for bevacizumab- containing regimens), radiotherapy, or surgical procedure with resolution of all treatment-related toxicity to NCI CTCAE Version 4.0 grade ≤1 (or tolerable grade 2) or back to baseline except for alopecia or hypothyroidism.
* Patients must have RECIST v1.1 measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as > or = to 20 mm with conventional techniques or as > or = to 10 mm with spiral CT scan.
* Patients must have documentation of a new or progressive lesion on a radiologic imaging study performed within 6 months prior to study enrollment (progression of disease over any interval is allowed) and/or new/worsening disease related symptoms. Note: This assessment will be performed by the treating investigator. Evidence of progression by RECIST criteria is not required.
* Patients must have archival tissue from the primary tumor or metastases available for correlative studies. Either a paraffin block or twenty unstained slides containing 5μm sections are acceptable. If twenty slides are not available, a lesser amount may be acceptable after discussion with the study Principal Investigator, Dr. Alan L. Ho.
* Male or female, age > or = to 18 years.
* ECOG performance status < or = to 2 (Karnofsky > or = to 60%, see Appendix A).
* Life expectancy of ≥ 12 weeks.

Adequate organ function as defined by the following criteria:

* absolute neutrophil count (ANC) > 1000 cells/mm3
* platelets > or = to 75,000 cells/mm3
* Hemoglobin > or = to 9.0 g/dL
* AST and ALT < or = to 2.5 x upper limit of normal (ULN), unless there are liver metastases in which case AST and ALT < 5.0 x ULN
* Total bilirubin < or = to 1.5 x ULN
* Serum creatinine < or = to 1.5 x ULN or calculated creatinine clearance > or = to 60 ml/min
* Urinary protein < 2+ by urine dipstick. If dipstick is > or = to 2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is < 2 g per 24 hours.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months after discontinuing study treatment.

Exclusion Criteria:

* Major surgery < 2 weeks or radiation therapy < 2 weeks of starting the study treatment.
* Gastrointestinal abnormalities including:

  * inability to take oral medication;
  * malabsorption syndromes.
* Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (i.e., grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine)
* Current use or anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (i.e., carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort)
* Requirement for anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
* Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Female patients who are pregnant or lactating.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan L. Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 03-15-2012, Protocol Closed to Accrual 08-27-2013, Primary Completion Date 08-25-2016, Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | AG-013736 (AXITINIB)
Started | 33
First Stage | 18
Second Stage | 15
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AG-013736 (AXITINIB)
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Best overall response rate documented by RECIST v1.1 criteria of patients with progressive, recurrent/metastatic ACC treated with axitinib. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions
Time Frame: 2 years
Population: One patient enrolled in the second stage was determined to be ineligible and was replaced after two doses. This patient was considered evaluable for Best Overall Response, but not for Progression Free Survival.
Measure: Count of Participants; unit: Participants
Arm/Group | AG-013736 (AXITINIB)
Number analyzed (Participants) | 33
Participants
  Complete Response | 0
  Partial Response | 3
  Stable Disease | 25
  Progressive Disease | 4
  Non-evaluable | 1

2. Secondary Outcome: Median Progression-free Survival (PFS).
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions"
Time Frame: 2 years
Population: One patient enrolled in the second stage was determined to be ineligible and was replaced after two doses. This patient was considered evaluable for Best Overall Response, but not Progression Free Survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-013736 (AXITINIB)
Number analyzed (Participants) | 32
months | 5.7 [5.3 to 9.1]

3. Secondary Outcome: MYB Immunohistochemistry (IHC)
Time Frame: 2 years
Population: MYB immunohistochemistry (IHC) was carried out on tumors from 33 patients. MYB quantification was assessed as: 2+ for strong staining in >50% of cancer cells, 1+ for weak or strong staining in <50% of the cells and 0 for <5% staining.
Measure: Count of Participants; unit: Participants
Arm/Group | AG-013736 (AXITINIB)
Number analyzed (Participants) | 33
Participants
  MYB IHC Testing Not Done | 7
  MYB IHC Score 0 | 13
  MYB IHC Score +1 | 8
  MYB IHC Score +2 | 5

4. Secondary Outcome: Number of Participants With Next Generation Sequencing (NGS)
Description: Next generation sequencing the t(6;9) translocation (MYBNFIB gene product) status will be analyzed by Fluorescent In-Situ Hybridization (FISH) assay and correlated to clinical response. The number of participants with NGS will be recorded.
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AG-013736 (AXITINIB)
Number analyzed (Participants) | 33
Participants
  No NGS sequencing | 22
  NGS sequencing | 11

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Toxicity will be graded using Common Terminology Criteria for Adverse Events version 4.0 (CTCAE version 4.0).
Arm/Group | AG-013736 (AXITINIB)
All-Cause Mortality (participants affected / at risk) | 25/33
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (AXITINIB) (N=33)
Alanine aminotransferase increased (Investigations) | 2
Alkaline Phosphatase Increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 3
Confusion (Psychiatric disorders) | 1
Corneal Ulcer (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Death NOS (General disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infections and infestations - Other (Infections and infestations) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Seizure (Nervous system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (AXITINIB) (N=33)
Hypertension (Vascular disorders) | 32
Fatigue (General disorders) | 30
Anorexia (Metabolism and nutrition disorders) | 18
Diarrhea (Gastrointestinal disorders) | 18
Hyperglycemia (Metabolism and nutrition disorders) | 18
Weight loss (Investigations) | 18
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Alanine aminotransferase increased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 14
Oral pain (Gastrointestinal disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Mucositis oral (Gastrointestinal disorders) | 12
Anemia (Blood and lymphatic system disorders) | 11
Aspartate aminotransferase increased (Investigations) | 9
Platelet count decreased (Investigations) | 9
White blood cell decreased (Investigations) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Dysphagia (Gastrointestinal disorders) | 8
Blood bilirubin increased (Investigations) | 7
Constipation (Gastrointestinal disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7
Hypothyroidism (Endocrine disorders) | 7
Hemoglobin increased (Investigations) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Headache (Nervous system disorders) | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Pain (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Proteinuria (Renal and urinary disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Serum amylase increased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes